CLINICAL TRIAL: NCT03783676
Title: Does Precise Delivery of Remifentanil Decrease Coughing at Emergence From Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Elie Sarraf, Principal Investigator, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 18-0415
Record Dates: First submitted 2018-12-15; First posted 2018-12-21 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Cough
Keywords: extubation
MeSH Terms: conditions — Cough | interventions — Remifentanil; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Remifentanil group (Experimental): Will receive remifentanil bolus and infusion guided by an algorithm
  Interventions: Drug: Remifentanil
- Control group (Placebo Comparator): Will receive normal saline bolus and infusion guided by the remifentanil algorithm
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Remifentanil — Receive remifentanil bolus and infusion guided by an algorithm.
  Arms: Remifentanil group
Drug: Normal saline — Receive normal saline bolus and infusion guided by the remifentanil algorithm.
  Arms: Control group

SUMMARY:
The investigators want to find a way to reduce or stop patients from coughing at the end of surgery when the breathing tube is taken out. The breathing tube is removed when the participants are waking up from anesthesia, and are at the point when the participants can breathe on your own. In most types of surgery, coughing at this point is common, and does not affect the participants very much, if at all. But for surgery involving the eye or the head and neck, coughing right after surgery can cause bleeding at the site of surgery.

This study will use a short-acting pain drug called remifentanil at the end of surgery to prevent coughing. The investigators will give the participants this medicine for 5 to 30 minutes. The point of the study is to test if using a simple computer program to guide precise delivery of how much of the drug is given to the participants is effective at reducing or preventing coughing.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 80
2. ASA of 1-3
3. Undergoing any of the following elective cases:

   1. thyroidectomy (partial or complete)
   2. parathyroidectomy
   3. ophthalmological surgery
4. Will require endotracheal intubation.

Exclusion Criteria:

1. Lean Body Mass < 20 kg,
2. BMI > 45
3. Presence of pulmonary dysfunction
4. Any history of anaphylaxis to remifentanil
5. Requiring the use of total intravenous anesthesia.
6. Per the discretion of the anesthesia provider

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of cough | Measured from surgical end time to patient transfer out of room, approximetly 30 minutes and up to 45 minutes
  Notes presence of cough during emergence

SECONDARY OUTCOMES:
Coughing grade | Measured from surgical end time to patient transfer out of room, approximetly 30 minutes
  Ranks severity of cough during emergence: cough was graded according to the following scoring guidelines: 0=no cough, 1=slight cough, cough without obvious contraction of the abdomen, 2=moderate cough, strong and sudden contraction of the abdomen lasting for less than 5 seconds and 3=severe cough, strong and sudden contraction of the abdomen sustained for more than 5 seconds.
Extubation time | Measured from termination of the anesthetic to extubation, approximetly 5 minutes and up to 30 minutes
  Time between the termination of the anesthetic and extubation
Time to recovery | Measured from extubation to purposeful movement, approximetly 5 minutes and up to 30 minutes
  Time between extubation and the ability to perform purposeful movement

CONTACTS AND LOCATIONS:
Overall Officials: Elie Sarraf, MD.CM., Principal Investigator — Resident

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Informed Consent Form (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03783676/ICF_000.pdf
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03783676/Prot_001.pdf